CLINICAL TRIAL: NCT02274324
Title: Dietary Modifications Effect on Continuous LCIG Infusion Outcomes in Patients With Advanced Parkinson's Disease
Brief Title: Dietary Modifications Effect on Continuous LCIG Infusion Outcomes in Patients With Advanced Parkinson&Apos;s Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dr. Oren Cohen, Dr, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1310-14-SMC
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Parkinson Disease
Keywords: parkinson; duodopa; diet; proteins; amino acids
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PD patients- Diet B first (Active Comparator): Patients treated with Duodopa at least three months and are stable on medical therapy. The intervention cosists of Dietary Change. Patients that will be randomized to this group will start diet B and then crossover to diet C.
  Interventions: Dietary Supplement: different diets
- PD patients- Diet C first (Active Comparator): Patients treated with Duodopa at least three months and are stable on medical therapy. The intervention cosists of Dietary Change. Patients that will be randomized to this group will start diet C and then crossover to diet B.
  Interventions: Dietary Supplement: different diets

INTERVENTIONS:
Dietary Supplement: different diets — 3 different diets: A\B\C

SUMMARY:
To evaluate the role of dietary modifications of 3 different diets on clinical outcomes in patients with PD treated with Duodopa®. This is in search for an optimal diet that will accompany Duodopa® treatment and will optimize effect on fluctuations and dyskinesias and thus improve motor function and quality of life.

DETAILED DESCRIPTION:
A prospective single-blind-crossover study in patients with PD regularly treated with Duodopa® (LICG) in which three different diets will be given. Diet A: Low fat western diet - traditional low-fat Western diet; a normal diet according to the recommendations of health organizations in which proteins consumed throughout the day, high-protein meal at noon and in the evening.

Diet B: Equal protein redistribution diet (EPRD) - proteins consumption is controlled and equally distributed over six meals throughout the day to minimize motor fluctuations.

Diet C: Protein redistribution diet (PRD) in which proteins are consumed in the morning prior to connection to the pump and in the evening after disconnecting from the . Carbohydrates and fats will be consumed during the day.

Following recruitment and study initiation patients will consume diet A for 3 weeks. Patients will then be randomized into either diet B or diet C for 3 additional weeks. At completion of this period patients will consume diet A for 2 weeks ("wash-out" period) and will then be "crosseovered" to get the third diet (B or C).

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Duodopa at least three months and are stable on medical therapy
* Patients should be not demented, able to fill diaries and to sign an informed consent

Exclusion Criteria:

* Severe dementia
* Inability to fill out diaries
* Unstable mediated condition
* Chronic renal failure

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
quality of life | 4 months
  CGI, PDQ-39
dyskinesias | 4 months
  AIMS

SECONDARY OUTCOMES:
fluctuations | 4 months
  questioners regarding "off" time
motor function | 4 months
  UPDRS

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Hassin, Dr, Study Director — Sheba Medical Center; Oren Cohen, Dr, Principal Investigator — Sheba Medical Center